CLINICAL TRIAL: NCT06872203
Title: LFP Sensing From Directional Leads and Associated Clinical Outcomes in the Acute Clinical Setting
Brief Title: LFP Sensing From Directional Leads in the Acute Clinical Setting
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 21-4938
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease, Idiopathic; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PD patient: PD patient after receiving a Medtronic DBS implant.
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Deep Brain Stimulation programming

SUMMARY:
This study plans to learn more about the optimal way to program the Medtronic Deep Brain Stimulation system in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
The investigators will conduct a prospective study in patients with Parkinson's disease (PD) implanted with standard of care, subthalamic nucleus (STN) deep brain stimulation (DBS) electrodes, to test whether monopolar sensing of the maximal power in the beta frequency range (in STN) predicts the optimal therapeutic stimulation setting for alleviation of PD motor symptoms. Participants in this study will have been implanted with a Medtronic DBS system consisting of a PerceptTM PC neurostimulator (battery) and SenSight™ DBS leads (implanted electrodes) with BrainSenseTM technology. The DBS surgery is a standard of care procedure, and no alteration of the surgical plan will occur for research purposes . The ranked response between the clinical profile (therapeutic benefit and adverse effects) and beta power will be compared for all electrical contacts on the implanted electrode. Additional analysis of monopolar sensing compared to differential bipolar sensing, location/distance and volume of neural activation (VNA) of optimal contacts identified by beta power or therapeutic window will be estimated with respect to the STN.

Aim 1- Determine whether monopolar sensing of beta power, in the outpatient clinic setting, will predict the optimal therapeutic contact for electrical stimulation of the STN.

Aim 2 - Long Term Follow Up (>12 months) of the same consented study participants to determine the stability of the beta power to determine the optimal contact for therapeutic stimulation.

ELIGIBILITY:
Inclusion Criteria: Parkinson's Disease, scheduled to undergo bilateral subthalamic nucleus (STN) Deep Brain Stimulation (DBS) surgery at the University of Colorado Hospital, chosen to have a Medtronic Deep Brain Stimulation system implanted (Percept™ battery & SenSight™ electrode). Parkinson's Disease causes upper extremity bradykinesia (slowness of movement) with a MDS-UPDRS1score of 2 or higher when you are off your PD medications.

-

Exclusion Criteria: Dementia or other psychological disorders that precludes consent to participate. Inability to follow testing procedures as determined by the study doctor. Inability to be OFF medication for study visits. Existing implanted Deep Brain Stimulation system or implanted cardiac device. Unilateral Medtronic DBS system, or programming not occurring at the University of Colorado Hospital.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients undergoing implantation of Medtronic DBS system; Sensight(TM) lead and Percept (TM) battery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To compare beta frequency power to the TW of each contact. | 2 study visits of 4 hours each, one week apart.
  Contacts will be ranked from highest to lowest in beta frequency power and compared to the rankings of the TW from largest to least. It is hypothesized that there will NOT be a statistically significant difference between the ranks for beta power and TW. This would indicate that the contact with the highest beta frequency power also had the largest TW and the converse also being evident.

CONTACTS AND LOCATIONS:
Overall Officials: John A Thompson, PhD, Study Director — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No